CLINICAL TRIAL: NCT05757037
Title: Laser Acupuncture for Treatment of Female Patients With Irritable Bowel Syndrome:RCT
Brief Title: Laser Acupuncture on Irritable Bowel Syndrome in Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ahmed, PRINCIPAL INVESTIGATOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T/WH/2/2023/31
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture group (Experimental): The participants in this group will receive low level laser therapy 3 times weekly for 4 weeks. A diode laser emitter with a 650 nm wavelength, an average power of 30 mW, and a 0.15 cm2 spot size, with continuous wave, and exposure of 90 s per acupuncture point had been used in the current study at each of the following acupoints: : ST25, ST37 , LI11 , BL60 , and BL25 Also, participants will recieve received behavioral therapy advice: Sitting on the toilet for 10-15 min after breakfast and after dinner and maintaining the same bathroom schedule every day, sitting in the correct position on the toilet (leaning forward while resting forearms on thighs, raising both feet on a small block (like a step stool) with feet apart, relax and lower the shoulders, and do not suppress urges to defecate and relax stomach muscles). Dietary modifications include a high-fiber diet, fruits, vegetables, whole grain, dairy, and wheat
  Interventions: Device: laser acupuncture
- Sham laser acupuncture (Sham Comparator): The participants in the control group will receive sham laser acupuncture treatment, without any laser output. The participants are unable to recognize whether they are being treated or not because laser acupuncture is a low-intensity and non-thermal laser irradiation.
  Also, participants will receive behavioral therapy advice.
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — a gallium aluminum arsenide LaserPen (maximal power, 150 mW; wavelength, 810 nm; area of probe, 0.03 cm2; power density, 5W/cm2; pulsed wave; and Bahr frequencies [B1: 599.5Hz, B2: 1199Hz, B3: 2398Hz, B4: 4776Hz, B5: 9552 Hz, B6: 19,104Hz, and B7: 38,208Hz].

SUMMARY:
The aim of the study to investigate effect of laser acupuncture on constipation predominant irritable bowel syndrome in female patients

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common chronic functional gastrointestinal disorder characterized by recurrent abdominal pain and/or bloating related to defecation without reliable biological markers . IBS is associated with substantial burden, such as higher levels of anxiety, lost productivity at work, work absenteeism (Pimentel, 2018). IBS has a strong predominance in women IBS-C includes a wide range of symptoms, and its pathophysiology is complex and not fully understood. Visceral hypersensitivity and delayed gut transit are recognized as major pathophysiological mechanisms in IBS-C. Visceral hypersensitivity may account for symptoms of abdominal pain, bloating, and discomfort. Delayed gut transit causes constipation The unsatisfactory treatment responses and adverse effects associated with pharmacologic therapies have resulted in a higher demand for alternative therapies Acupoints and manipulations are the same in both the experimental and the control groups. The participants in the control group will receive sham laser acupuncture treatment, without any laser output, while the participants in the experimental group will sequentially receive 0.375J of energy at each of the following acupoints: Baihui (GV20), Yintang (GV29), Taichong (LR3), Zusanli (ST36), Sanyinjiao (SP6), Tianshu (ST25), and Shangjuxu (ST37) acupoint .Using a gallium aluminum arsenide LaserPen (maximal power, 150 mW; wavelength, 810 nm; area of probe, 0.03 cm2; power density, 5W/cm2; pulsed wave; and Bahr frequencies [B1: 599.5Hz, B2: 1199Hz, B3: 2398Hz, B4: 4776Hz, B5: 9552 Hz, B6: 19,104Hz, and B7: 38,208Hz]. The laser treatment will be applied to each point for 5 seconds, to deliver a total treatment dose of 4.5J/cm2 . intervention will be 3t/ week for 6 weeks in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All participants will meet diagnostic criteria (Rome IV) for IBS-C
* Their age will range from 20-35 years old
* Their body mass index (BMI) will range from >18.5kg/m2 and <29.9kg/m2

Exclusion Criteria:

* Taking medications known to cause constipation
* Any organic diseases that might induce constipation such as colorectal cancer, metabolic disorders, multiple sclerosis, or neurological disorders
* Organic diseases of the small or large intestine such as ulcerative colitis and Crohn's disease
* A history of gastrointestinal surgery (other than appendectomy or cholecystectomy)
* Mechanical obstruction
* Serious concomitant disease of the heart, liver, or kidney or diabetes
* Pregnant or lactating women
* Severe psychiatric disorders
* Knowledgeable of acupoints and meridians that might unblind the treatment.

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The number of complete spontaneous bowel movement (CSBMs) per week (Zhihui et al., 2022) | 6 weeks
Irritable Bowel Syndrome Severity Score (IBS-SSS) | 6 weeks

SECONDARY OUTCOMES:
IBS Quality of Life (IBS-QOL) (Andrae et al., 2013) | 6 weeks
Visceral Sensitivity Index (VSI) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt , Giza, Giza, Egypt